CLINICAL TRIAL: NCT07308977
Title: Factors Affecting the Practice of Assisted Vaginal Birth in Three Tertiary Level Hospitals in Egypt. A Cross-Sectional Study
Brief Title: Practice of Assisted Vaginal Birth in Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Elmaraghy, Assistant professor of Obstetrics and Gynecology, Ain Shams Maternity Hospital
Other Study IDs: 20
Record Dates: First submitted 2025-12-04; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Vaginal Delivery
Keywords: Assisted vaginal delivery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey using a questionnaire. — This cross-sectional study aims to identify the obstacles preventing an increase in AVB performance in Egypt. Obstetricians from three tertiary care centers in Egypt will be invited to participate in this Online web-based survey over the study period. The questions in this survey are included in 5 sections; demographics, workload and AVB practice, obstetrician-related factors, service provision factors, and what changes could be implemented to increase the rate of uptake of AVB by Egyptian obstetricians. The link to the survey will be sent to the study participants, and the data will be collected for analysis

SUMMARY:
In Egypt, the proportion of CSs has been steadily increasing in recent years and has reached an alarming level. According to data from the Royal College of Obstetricians and Gynaecologists (RCOG), approximately 6% of caesarean sections (CS) are performed on average because of inadequate supervision from junior staff members or a lack of training, particularly during the critical decision-making phase of this second stage. The unfamiliarity and lack of experience with operative vaginal delivery is a major cause for the rise in the rate of second stage caesarean section. This survey targets obstetricians with different levels of experience to find practical solutions to increase the rate of assisted vaginal delivery which subsequently will decrease the rate of second stage CS.

DETAILED DESCRIPTION:
Egypt is a populous African country with a population of about 102 million people in 2020. Egypt has the highest cesarean section (CS) rate in the Middle East, which has increased from 20% in 2005 to 52% in 2014. Globally, the estimated number of births by Cesarean section (CS) increased from 16 million (12%) in 2000 to 29.1 million (21%) in 2015. Furthermore, during the same period, several studies have demonstrated a remarkable increase in the rate of second-stage cesarean section.

Whereas forceps-assisted vaginal delivery represented 38% of deliveries in rural areas of Egypt, in the United States, operative vaginal delivery in the form of either forceps-assisted vaginal delivery (FAVD) or ventouse-assisted vaginal delivery (VAVD) has declined remarkably since 1990. The utilization of operative vaginal delivery in live births decreased from 9.0% in 1990 to 3.1% in 2016. During the same period, the percentage of VAVD deliveries fell from 3.9 to 2.6%, and FAVD from 5.1 to just 0.5%. The declining rate of assisted vaginal delivery contributed to the rise in the cesarean section rate from 22.7% in 1990 to 31.9% in 2016.

The performance of AVB by physicians with a high level of experience and certified training courses should be considered a safe alternative to second-stage cesarean section. This does not only depend on the physician, but it also depends on the patient's preference. In this survey, the investigators explore Egyptian obstetricians 'attitudes and perceptions on AVB.

ELIGIBILITY:
Inclusion Criteria:

* Obstetricians with at least 3 years of experience in practicing obstetrics
* Obstetricians with their primary health care facility being one of the three Tertiary centres, Ain Shams University Maternity Hospital, El Hussein University Hospital, and El Kasr Alaini Hospital

Exclusion Criteria:

-

Ages: 28 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obstetricians from three tertiary maternity hospitals in Cairo, Egypt. The three hospitals are Ain Shams University Maternity Hospital, El Hussein University Hospital, and El Kasr Alaini Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Obstacles preventing the increase in the performance of assisted vaginal birth in Egypt by a questionnaire directed to obstetricians in three maternity tertiary centers in Cairo, Egypt | through the study completion, an average of 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Alaa S Elsewafy, M.D.,, Study Chair — Faculty of Medicine - Ain Shams university; Mohamed A Haroun, Principal Investigator — Faculty of Medicine - Modern University for Technology and Information; Ahmed M Sweidan, Study Chair — Faculty of Medicine - Suez University

REFERENCES:
- [Background] Obstetric care consensus no. 1: safe prevention of the primary cesarean delivery. Obstet Gynecol. 2014 Mar;123(3):693-711. doi: 10.1097/01.AOG.0000444441.04111.1d. PMID 24553167
- [Background] Becker DA, Blanchard CT, Szychowski JM, Rogers SL, Brumfield CG, Subramaniam A. Resident Operative Vaginal Delivery Volume after Educational Curriculum Implementation. Am J Perinatol. 2020 Nov;37(13):1296-1300. doi: 10.1055/s-0040-1710543. Epub 2020 May 26. PMID 32455468
- [Background] Darmstadt GL, Hussein MH, Winch PJ, Haws RA, Gipson R, Santosham M. Practices of rural Egyptian birth attendants during the antenatal, intrapartum and early neonatal periods. J Health Popul Nutr. 2008 Mar;26(1):36-45. PMID 18637526
- [Background] Banerjee A, Al-Dabbach Z, Bredaki FE, Casagrandi D, Tetteh A, Greenwold N, Ivan M, Jurkovic D, David AL, Napolitano R. Reproducibility of assessment of full-dilatation Cesarean section scar in women undergoing second-trimester screening for preterm birth. Ultrasound Obstet Gynecol. 2022 Sep;60(3):396-403. doi: 10.1002/uog.26027. PMID 35809243
- [Background] Jadoon B, Assar TM, Nucier AAAR, Raziq HEA, Abd El-Azym Saad AS, Megahed Amer W. Analysis of the caesarean section rate using the 10-Group Robson classification at Benha University Hospital, Egypt. Women Birth. 2020 Mar;33(2):e105-e110. doi: 10.1016/j.wombi.2019.03.009. Epub 2019 Apr 13. PMID 30987799
- [Background] Fasseeh A, ElEzbawy B, Adly W, ElShahawy R, George M, Abaza S, ElShalakani A, Kalo Z. Healthcare financing in Egypt: a systematic literature review. J Egypt Public Health Assoc. 2022 Jan 7;97(1):1. doi: 10.1186/s42506-021-00089-8. PMID 34994859